CLINICAL TRIAL: NCT00899184
Title: Assessment of SNP Genotypes in Men With Prostate Cancer
Brief Title: DNA Changes in Patients With Prostate Cancer
Status: Completed | Type: Observational
Sponsor: ECOG-ACRIN Cancer Research Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: Eastern Cooperative Oncology Group (Network)
Other Study IDs: CDR0000492784; ECOG-E1Y97T1; ECOG-O00PCONS01
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2017-05-19 (Actual); Status verified 2017-05

CONDITIONS: Prostate Cancer
Keywords: recurrent prostate cancer; stage IV prostate cancer; stage I prostate cancer; stage IIB prostate cancer; stage IIA prostate cancer; stage III prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Amplified Fragment Length Polymorphism Analysis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective

INTERVENTIONS:
Genetic: polymorphism analysis
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Collecting and storing samples of blood from patients and their brothers with cancer to study in the laboratory may help doctors learn more about changes that may occur in DNA and identify biomarkers related to cancer.

PURPOSE: This laboratory study is looking at changes in DNA in patients and their brothers with prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the frequency of single nucleotide polymorphism (SNP) genotypes in patients with prostate cancer, their affected siblings, and an unaffected healthy population (control).
* Determine the age of onset of prostate cancer in affected probands and affected siblings.
* Determine the penetrance or likelihood that given SNPs will result in disease in affected siblings based upon Mendelian genetics.
* Determine the odds ratio of developing prostate cancer in the presence of SNPs.
* Determine SNP genotypes in patients enrolled on ECOG-E3805, a prostate phase III study enrolling men with D2 prostate cancer treated with androgen-ablation therapy alone or androgen-ablation therapy with chemotherapy, and correlate them with disease progression (i.e., androgen independence).

OUTLINE: This is an open-label, multicenter study. Patients are stratified according to ethnicity, age at diagnosis, and Gleason score.

Patients, their affected siblings, and healthy participants (controls) undergo collection of blood samples. Genomic DNA is extracted from whole blood and sequenced for single nucleotide polymorphisms (SNPs) in Akt and mdm-2 genes. SNP data is correlated with clinical and biographical data.

PROJECTED ACCRUAL: A total of 500 patients (250 probands and 250 siblings) and 146 healthy participants (controls) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Meets one of the following criteria:

  * Patient or sibling diagnosed with prostate cancer
  * Cancer-free participant (healthy control)
* Whole blood sample available

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Ages: 18 Years to 120 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 646 (Actual)
Dates: Start 2006-05-23 (Actual); Primary Completion 2007-05-30 (Actual); Study Completion 2007-05-30 (Actual)

PRIMARY OUTCOMES:
Frequency of single nucleotide polymorphism (SNP) genotypes | 1 month
Age of onset of prostate cancer in patients and their affected siblings | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Kim M. Hirshfield, MD, PhD, Study Chair — Rutgers Cancer Institute of New Jersey